CLINICAL TRIAL: NCT02653508
Title: Evaluating the Efficacy of the Feeding Exercise Trial in Adolescents (FETA Project) in Central Greece
Acronym: FETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Hadjichristodoulou Christos, Professor of Hygiene and Epidemiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: obesity1uth
Record Dates: First submitted 2015-12-17; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: BMI: Body Mass Index; obesity; adolescents; overweight; CI:confidence interval; CDC: Center Disease Control
MeSH Terms: conditions — Obesity; Overweight | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diet and Activity (Experimental): 60 overweight and obese adolescents aged 13-15 years old took part in the clinical trial and remained at the end of the 3 months intervention program and also at the 6 months follow up. The activity intervention included a 45 minutes, three-day per week supervised training programme, while the nutritional education comprised of a supplementary 15 minutes of group-based sessions that could be also attended by the parents. All adolescents were assessed for anthropometric measures, fitness and activity and family habits along with their parents.
  Interventions: Behavioral: Diet and Activity
- Activity (Experimental): 60 overweight and obese adolescents aged 13-15 years old took part in the clinical trial and remained at the end of the 3 months intervention program and also at the 6 months follow up. The activity intervention included a 45 minutes, three-day per week supervised training programme, that could be also attended by the parents. All adolescents were assessed for anthropometric measures, fitness and activity and family habits along with their parents.
  Interventions: Behavioral: Activity
- Control (No Intervention): 61 overweight and obese adolescents aged 13-15 years old were the control group of the clinical trial and remained at the end of the 3 months intervention program and also at the 6 months follow up. All adolescents were assessed for anthropometric measures, fitness and activity and family habits along with their parents.

INTERVENTIONS:
Behavioral: Diet and Activity — During all the following meetings, before the initiation of the training sessions, 10 to 15 minutes were devoted to an interactive discussion with participants on food pyramid, food choices, food labels, food preparation and cooking, eating habits, regular meals, controlling environments that stimulate overeating. All adolescents participated in a three-day per week training programme (45 minutes per training session). Many activities were delivered as games in order to encourage enthusiasm and participation. Endurance type activities accounted for most of the time spent in training (about 50% team sports and 50% running games), with attention to coordination and flexibility skills.
  Arms: Diet and Activity
Behavioral: Activity — All adolescents participated in a three-day per week training programme (45 minutes per training session). Training was directed by a professional teacher of physical education in a public training centre. The training program was designed according to the type and intensity of exercise that school children normally perform. Many activities were delivered as games in order to encourage enthusiasm and participation. Endurance type activities accounted for most of the time spent in training (about 50% team sports and 50% running games), with attention to coordination and flexibility skills. In order to encourage adolescents' behaviour change, they were instructed to add an extra 30-45 minutes of walking or other sport activity of their preference at least once a week and to reduce inactivity
  Arms: Activity

SUMMARY:
The Feeding-Exercise Trial in Adolescents (FETA) was a randomised controlled intervention study designed to promote healthy weight in overweigh and obese adolescents through a professional-delivered, community-based program with active parents' involvement, focused on supervised physical activity and structured nutritional education. The aim of FETA was to test the efficacy of two intervention groups- physical activity in isolation and combination of physical activity with provision of dietary information- for improving overweight and obesity in adolescents. Our primary hypothesis was that a combined program would be more efficacious than activity in isolation and that activity alone would also be effective compared to control group in improving adiposity profiles in overweight and obese adolescents as well as family activity and feeding habits.

DETAILED DESCRIPTION:
Study design:

All students from the 15 public middle schools in the city of Larissa in central Greece were invited to measure their weight and height, in order to calculate their Body Mass Index (BMI). All the overweight or obese students were invited to take part in the study. The participation was free of charge for the children. Parents were informed about the purposes of the project and were asked to provide written informed consent for participation. The study's protocol was approved by the ethics committee of the Medical Department of the University of Thessaly.

One hundred eighty one adolescents were enrolled and randomized in the three groups of the study, by the same professional teacher of physical education who conducted the program. One hundred fifty remained the end of the program and the 6-months follow up and were included in the analysis. None of the subjects had an organic cause for his/her obesity and none received any medication, which would interfere with growth or weight control (e.g. corticosteroids, thyroid hormone).

Intervention:

The FETA project involved one control and two intervention groups: a Physical Activity Skill Development Program (Activity) and a combination of a Dietary Information and a Physical Activity Skill Development Program (Diet and Activity).

Physical Activity Skill Development Program:

All adolescents participated in a three-day per week training programme (45 minutes per training session). Training was directed by a professional teacher of physical education in a public training centre. The training program was designed according to the type and intensity of exercise that school children normally perform. Many activities were delivered as games in order to encourage enthusiasm and participation. Endurance type activities accounted for most of the time spent in training (about 50% team sports and 50% running games), with attention to coordination and flexibility skills. In order to encourage adolescents' behaviour change, they were instructed to add an extra 30-45 minutes of walking or other sport activity of their preference at least once a week and to reduce inactivity (discouraging television watching and playing video games and encouraging the use of stairs instead of lifts and playing outdoors).

Structured nutrition education:

Additionally, to the training sessions, the participants of the combined intervention attended a structure nutrition educational program. In the introductory meeting (45-60 minutes) general information was presented about the reasons behind childhood obesity, dietary and cooking habits and the motivation for weight loss in an effort to involve the whole family in the ''battle'' against obesity. During all the following meetings, before the initiation of the training sessions, 10 to 15 minutes were devoted to an interactive discussion with participants on food pyramid, food choices, food labels, food preparation and cooking, eating habits, regular meals, controlling environments that stimulate overeating. The topics discussed were given to the adolescents in the form of a printed notebook, while parents were also invited to attend these sessions. The discussions were led by the same person who performed the training session.

Outcome measures:

All the outcomes measures were taken at baseline and every month until the end of the sixth month, when the 3-month follow up period after the intervention ended.

1. Anthropometric measurements:

   Students were weighed on a digital scale twice and the average was recorded. Participants removed shoes and jackets before heights and weights were measured. Participants' heights were measured using a metric measuring tape affixed on the wall. Body weight and height were measured using the same instruments, at the same place and day of the week, before the start of the day's program. Non-extensible steel tapes were used to assess waist circumference, which was measured at the level of the mid point between the lower costal border and the iliac crest. All the anthropometric measures were conducted using the International Society for the Advancement of Kin anthropometry procedures. BMI was determined according to the following formula: BMI= [weight/height2]. We used the cut off points for the BMI in childhood presented by Cole et al in order to allow international comparisons with our findings in the prevalence of overweight and obesity. Pulses per minute were measured using an automated blood pressure monitor under standardised procedures.
2. Fitness assessment:

   Pre- and post- intervention evaluations (at 3 and 6 months) of physical fitness were based on the EUROFIT Tests Protocol designed by the Committee of Experts on Sports Research that has been used in several European countries. The 50m sprint Run Test that was used is a test for the evaluation of speed.
3. Family Eating and Activity Habits Questionnaire:

The modified version of the Family Eating and Activity Habits Questionnaire (FEAHQ) was completed by parents and adolescents. FEAHQ is divided into four subscales: activity level (4 items), stimulus exposure (8 items), eating related to hunger (4 items), and eating style (13 items).

Blinding:

The randomized adolescents in each group were not aware of the existence of the other two study groups. This was achievable by programming the attendance of each group at different hours, even on the same days. Moreover their parents were also unaware of the study's design. Finally, all the participants from each of the three groups- both adolescents and parents- were asked not to discuss their study experience until the completion of the follow up, at 6-months from the initiation of the study.

ELIGIBILITY:
Inclusion Criteria:

* None of the subjects had an organic cause for his/her obesity and
* none received any medication, which would interfere with growth or weight control (e.g. corticosteroids, thyroid hormone).

Exclusion Criteria:

* subjects who had an organic cause for his/her obesity
* subjects who received any medication, which would interfere with growth or weight control

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | change from baseline at 3 months intervention program
  Change in BMI (kg/m2)
Weight | change from baseline at 3 months intervention program
  Change in weight (kilograms)
Height | change from baseline at 3 months intervention program
  Change in height (meters)
Heart rate | change from baseline at 3 months intervention program
  Change in heart rate (beats per minute)
Blood Pressure | change from baseline at 3 months intervention program
  Change in Blood Pressure (mm Hg)
Waist circumference | change from baseline at 3 months intervention program
  Change in waist circumference (cm)
50m sprint Run Test | change from baseline at 3 months intervention program
  Change in 50m sprint Run Test (seconds)
Family Eating and Activity Habits | change from baseline at 3 months intervention program
  Change in <<Family Eating and Activity Habits>> (sum of the items)

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Change from Baseline at 6 months (follow up)
  Change in BMI (kg/m2)
Weight | Change from Baseline at 6 months (follow up)
  Change in weight (kilograms)
Height | Change from Baseline at 6 months (follow up)
  Change in height (meters)
Heart Rate | Change from Baseline at 6 months (follow up)
  Change in heart rate (beats per minute)
Blood Pressure | Change from Baseline at 6 months (follow up)
  Change in Blood Pressure (mm Hg)
Waist circumference | Change from Baseline at 6 months (follow up)
  Change in waist circumference (cm)
50m sprint Run Test | Change from Baseline at 6 months (follow up)
  Change in 50m sprint Run Test (seconds)
Family Eating and Activity Habits | Change from Baseline at 6 months (follow up)
  Change in <<Family Eating and Activity Habits>> (sum of the items)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Hadjichristodoulou, Professor, Study Director — Department of Hygiene and Epidemiology Medical School - University of Thessaly

IPD SHARING:
Plan to Share IPD: Yes
1. The data will be published
  2. The data will be given in the Ministry of Education and Religious Affairs, Sport and Culture of Greece

REFERENCES:
- [Result] Menghetti E, Strisciuglio P, Spagnolo A, Carletti M, Paciotti G, Muzzi G, Beltemacchi M, Concolino D, Strambi M, Rosano A. Hypertension and obesity in Italian school children: The role of diet, lifestyle and family history. Nutr Metab Cardiovasc Dis. 2015 Jun;25(6):602-7. doi: 10.1016/j.numecd.2015.02.009. Epub 2015 Mar 2. PMID 25858615
- [Result] Shikha D, Singla M, Walia R, Potter N, Umpaichitra V, Mercado A, Winer N. Ambulatory Blood Pressure Monitoring in Lean, Obese and Diabetic Children and Adolescents. Cardiorenal Med. 2015 Jun;5(3):183-90. doi: 10.1159/000381629. Epub 2015 Apr 30. PMID 26195970
- [Result] Okely AD, Collins CE, Morgan PJ, Jones RA, Warren JM, Cliff DP, Burrows TL, Colyvas K, Steele JR, Baur LA. Multi-site randomized controlled trial of a child-centered physical activity program, a parent-centered dietary-modification program, or both in overweight children: the HIKCUPS study. J Pediatr. 2010 Sep;157(3):388-94, 394.e1. doi: 10.1016/j.jpeds.2010.03.028. Epub 2010 May 6. PMID 20447648
- [Result] Hendrie GA, Brindal E, Corsini N, Gardner C, Baird D, Golley RK. Combined home and school obesity prevention interventions for children: what behavior change strategies and intervention characteristics are associated with effectiveness? Health Educ Behav. 2012 Apr;39(2):159-71. doi: 10.1177/1090198111420286. Epub 2011 Oct 7. PMID 21984691
- [Result] Manios Y, Moschandreas J, Hatzis C, Kafatos A. Evaluation of a health and nutrition education program in primary school children of Crete over a three-year period. Prev Med. 1999 Feb;28(2):149-59. doi: 10.1006/pmed.1998.0388. PMID 10048106